CLINICAL TRIAL: NCT01022944
Title: Prevalence of Mucosal Biofilm Formations in Adenoidectomy Specimens. A Case Control Study
Brief Title: Prevalence of Mucosal Biofilm Formations in Adenoidectomy Specimens
Acronym: BOLERO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P080605
Record Dates: First submitted 2009-09-30; First posted 2009-12-01 (Estimated); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Chronic Serous Otitis Media, Simple or Unspecified
Keywords: Serous otitis media; Biofilm; Adenoidectomy; Chronic otitis media
MeSH Terms: conditions — Charcot-Marie-Tooth disease, Type 1C; Otitis Media with Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 2 : (Other): Children without chronic middle ear effusion as a control group having adenoids removed for chronic obstruction.
  Interventions: Procedure: Without chronic middle ear effusion
- Group 1 (Other): Children with chronic middle ear effusion having adenoidectomy.
  Interventions: Procedure: With chronic middle ear effusion

INTERVENTIONS:
Procedure: With chronic middle ear effusion — Children with chronic middle ear effusion having adenoidectomy.
  Arms: Group 1
Procedure: Without chronic middle ear effusion — Children without chronic middle ear effusion as a control group having adenoids removed for chronic obstruction.
  Arms: Group 2 :

SUMMARY:
Rationale: Bacterial biofilms are defined as an assemblage of bacterial cells enclosed in a self-produced glycocalyx matrix. Adherence on surfaces, and resistance to both antibiotic treatments and host defenses are ones of the major clinical features of bacterial biofilms. Hence, biofilm formations represent a serious clinical problem: they persist in human tissues and play a role in a large number of chronic and resistant infections. It has been estimated that more than 65% of all human bacterial infections involve biofilms. Recently, the investigators have demonstrated the presence of mucosal bacterial biofilms in adenoid tissues removed during routine adenoidectomy. Bacterial biofilms were visualized using Confocal Laser Scanning Microscopy (CLSM) with a technique of double staining showing both the bacterial cells and the glycocalyx matrix. Although this study clearly established that adenoids tissues can harbour mucosal biofilms, the prevalence of 54% the investigators found suggested that some groups of children may contain more biofilm formations than others. In an effort to relate the findings of mucosal biofilm with the clinical presentation, the investigators have designed the present work to compare the prevalence of mucosal biofilms in adenoidectomy specimens in two groups: one group of children with chronic otitis media (COM) with effusion versus another group of children without any COM, having adenoids removed for chronic obstruction.

DETAILED DESCRIPTION:
The aim of this case-control study is to compare the prevalence of biofilms formations in adenoid tissues of children with COM versus a control group without any COM.

Design: This is a monocentric, prospective, unrandomized case-control study comparing the prevalence of biofilm formations in adenoid tissues of two groups.

Clinical research study without direct medical benefit: during routine adenoidectomy, specimens are not used and thrown away. This study do not modify the common management of included children.

Number of subjects required: A considered approach of simple size calculation have been made using a method proposed by MIETINEN for Mc NEMAR Chi2 test. Simple size N=104 will allow 80% power to detect different of 20% (absolute), considering a total percentage of discordance pair at 30 %.

Expected results: a higher prevalence (30% estimation) of biofilm formations in group 1 in comparison with that in group 2 would be the first clinical research study bringing understanding of the role of adenoid tissues by harboring mucosal biofilms in otitis prone children.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 and 2

  * obtained informed consent by both parents and child (if possible),
  * age > 18 months and <10 years
  * chronic serous otitis media lasting more than 3 months (group 1).
* Group 1 only:

  * chronic secretory otitis media
* Group 2 only:

  * hypertrophia adenoid vegetations without sinusal oropharyngeal infections

Exclusion criteria:

* No informed consent
* age < 18 months or > 10 years
* Eustachian tube dysfunction
* Immunodeficiency
* Tumor

Ages: 18 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2010-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of mucosal biofilm formations in adenoidectomy specimens analyzed using Confocal Laser Scanning Microscopy with double staining | at 2 years

SECONDARY OUTCOMES:
To build up a tissue bank of human tissue from adenoids and the middle ear for further bacterial identification | during the study

CONTACTS AND LOCATIONS:
Overall Officials: Romain KANIA, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital ROBERT DEBRE - ORL Pédiatrique, Paris, France